CLINICAL TRIAL: NCT02058979
Title: Pharmacokinetics of Bolus Versus Continuous Cefazolin Infusion in Patients Undergoing Major Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Principal Investigator, Bhiken I. Naik, MD, Assistant Professor, Anesthesiology, University of Virginia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17266
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Plasma Concentration of Antibiotics
MeSH Terms: interventions — Cefazolin; Infusion Pumps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOLUS INFUSION (Active Comparator): Bolus infusion of antibiotics
  Interventions: Drug: BOLUS INFUSION (Ancef)
- CONTINUOUS INFUSION (Experimental): Continuous infusion of antibiotics by way of infusion pump
  Interventions: Drug: CONTINUOUS INFUSION (Ancef)

INTERVENTIONS:
Drug: BOLUS INFUSION (Ancef) — Bolus Infusion of antibiotics
  Other Names: ANCEF Bolus Infusion of antibiotics
  Arms: BOLUS INFUSION
Drug: CONTINUOUS INFUSION (Ancef) — Continuous Infusion of ANCEF with infusion pump
  Other Names: Continuous Infusion of ANCEF with infusion pump
  Arms: CONTINUOUS INFUSION

SUMMARY:
Abstract The administration of an antibiotic preoperatively is an important intervention that helps to reduce the risk of post-operative health-care associated infections (HCAI). These include urinary tract, surgical site and blood stream infection. Based on the current Surgical Infection Prevention Project, (SCIP) recommendations, the choice of the antibiotic is based on the nature and site of the surgery and the presence of a β-lactam allergy (Table 1).

Currently, the antibiotic treatment for preventing surgical infections is administered as a single bolus an hour before surgery, and every four hours after the initial dose. This presents a concentration profile that has a high concentration after the bolus, but decays as the kidneys remove the antibiotics. In this present study, investigators would like to compare this traditional method of delivery to a constant infusion model that would sustain a constant level of antibiotics that is defined by the difference between the rate of infusion and rate of clearance.

DETAILED DESCRIPTION:
The current incidence of post-operative surgical infections varies between 6% for patients undergoing non-cardiac surgery to greater than 30% in high-risk surgery. 1 The administration of an antibiotic preoperatively is an important intervention that helps to reduce the risk of post-operative health-care associated infections (HCAI). These include urinary tract, surgical site and blood stream infection. Based on the current Surgical Infection Prevention Project, (SCIP) recommendations, the choice of the antibiotic is based on the nature and site of the surgery and the presence of a β-lactam allergy (Table 2). The antibiotic of choice for perioperative prophylaxis remains first and second generation cephalosporin. These drugs have a broad range of antimicrobial activity against common skin pathogens and have an excellent safety profile.

Based on current recommendations, the cephalosporin is administered 1 hour prior to incision.1 Timing is critical, as both early and late administration of the antibiotic is associated with an increase risk of HCAI. Additional doses of the cephalosporin are administered at pre-set intervals based on the duration of the surgery in an attempt to maintain antibiotic concentrations at a desired level.

Antibiotics can be classified into two broad classes, based on their bacterial killing characteristics. Antibiotics with concentration-dependent killing characteristics require a high ratio between the peak concentration and the minimum inhibitory concentration (MIC) of the pathogen, during the dosing interval. Therefore large infrequent doses of these antibiotics will result in optimal antibacterial activity.

In contrast β-lactam antibiotics, like cephalosporins, demonstrate time-dependent pharmacokinetics. This means that effective microbiological activity only occurs if the unbound (or free) plasma concentration of the drug is above the MIC for a specified time period. In infection models, bacteriostatic and bacteriocidical activity occurs when antibiotic concentrations are maintained above the MIC for 35-40% and 60-70% of the dosing interval respectively. However, in surgical prophylaxis, it is preferred that antibiotic concentrations are maintained above the MIC of the likely pathogen/s for the entire duration of the procedure. Therefore more frequent dosing or use of extended or continuous infusion of these drugs will better maintain the pharmacokinetic goals. Recent studies have shown that plasma levels of β-lactam antibiotics fall below the MIC 1-2 hours after the initial bolus dose in both normal and obese patients.2, 3 Even with appropriate re-dosing of the β-lactam antibiotic, there are times when the plasma concentration of the drug is below the MIC. The combination of sub-MIC plasma drug level and high bacteremic load can potentially increase the risk of developing a post-operative HCAI. It follows that to effectively prevent microbiological activity in the perioperative period the β-lactam antibiotic must remain above the MIC during the entire operative period. This is of particular importance in patients undergoing major abdominal surgery where the risk of perioperative surgical site infection (including superficial, deep and organ specific infection) is 13.1%. The aim of this study is to compare the pharmacokinetics of bolus and continuous cefazolin infusion during major abdominal surgery.

Hypothesis to be Tested Hypothesis A continuous infusion of cefazolin maintains the unbound plasma concentration above Minimum Inhibitory Concentration (MIC) for the duration of the operative procedure better than the traditional bolus administration at every four hours.

Specific Aims

1. Compare the pharmacokinetics of a bolus versus continuous cefazolin (Ansef) infusion in major surgery

A. Preliminary studies

There are 2 studies in the abdominal surgery population. The study by Troconiz et al studies the pharmacokinetics of a bolus dose of cefoxitin.3 The study by Suffoleta studied a postoperative continuous infusion in the postoperative colorectal group.4

B. Experimental design and methods (including data analysis)

Informed consent for the study will be obtained in the PETC (Pre-anesthesia Clinic) prior to surgery.

Induction and maintenance of anesthesia will be at the discretion of the attending anesthesiologist. Intraoperative analgesia will be provided at the discretion of the attending anesthesiologist and may include intravenous narcotics and/or intrathecal morphine.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Elective abdominal and orthopedic surgery
* A patent arterial line
* A patent IV line
* Must be able to read and speak English

Exclusion Criteria:

* Subjects unable to give informed consent.
* Allergy to cefazolin
* Cognitively Impared
* Prisoners
* Pregnant females (self reported)
* History of coagulopathy
* Subjects presenting for emergency abdominal surgery
* Creatinine clearance < 30 ml/min
* Received cefazolin within 72 hours prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of Antibiotics | 1 Day
  Plasma concentration of antibiotics during surgery

CONTACTS AND LOCATIONS:
Overall Officials: BHIKEN NAIK, M.B., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Suffoletta TJ, Jennings HR, Oh JJ, Stephens D, Poe KL. Continuous versus intermittent infusion of prophylactic cefoxitin after colorectal surgery: a pilot study. Pharmacotherapy. 2008 Sep;28(9):1133-9. doi: 10.1592/phco.28.9.1133. PMID 18752384
- [Background] Toma O, Suntrup P, Stefanescu A, London A, Mutch M, Kharasch E. Pharmacokinetics and tissue penetration of cefoxitin in obesity: implications for risk of surgical site infection. Anesth Analg. 2011 Oct;113(4):730-7. doi: 10.1213/ANE.0b013e31821fff74. Epub 2011 Jun 3. PMID 21642605
- [Background] Isla A, Troconiz IF, de Tejada IL, Vazquez S, Canut A, Lopez JM, Solinis MA, Rodriguez Gascon A. Population pharmacokinetics of prophylactic cefoxitin in patients undergoing colorectal surgery. Eur J Clin Pharmacol. 2012 May;68(5):735-45. doi: 10.1007/s00228-011-1206-1. Epub 2012 Jan 15. PMID 22246211
- [Background] Bratzler DW, Hunt DR. The surgical infection prevention and surgical care improvement projects: national initiatives to improve outcomes for patients having surgery. Clin Infect Dis. 2006 Aug 1;43(3):322-30. doi: 10.1086/505220. Epub 2006 Jun 16. PMID 16804848
- [Derived] Naik BI, Roger C, Ikeda K, Todorovic MS, Wallis SC, Lipman J, Roberts JA. Comparative total and unbound pharmacokinetics of cefazolin administered by bolus versus continuous infusion in patients undergoing major surgery: a randomized controlled trial. Br J Anaesth. 2017 Jun 1;118(6):876-882. doi: 10.1093/bja/aex026. PMID 28505360